CLINICAL TRIAL: NCT03763552
Title: Arthroscopic Midcarpal Wrist Arthrodesis: Clinical and Functional Outcomes
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH ID 2017-02003
Record Dates: First submitted 2018-09-10; First posted 2018-12-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Dislocation of Midcarpal Joint
Keywords: arthroscopy; wrist osteoarthrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: arthroscopic wrist arthrodesis — Cases of midcarpal wrist arthritis treated surgically with arthroscopic partial wrist fusion with cannulated screws

SUMMARY:
All cases of midcarpal wrist arthritis treated surgically with arthroscopic partial wrist fusion with cannulated screws from January 2015 to December 2017 will be reviewed.

The union rate and time to union will be recorded following the standard radiological postoperative control. Wrist assessments performed pre- and postoperative regarding strength, range of motion and pain will be analysed. Complications will be recorded as well.

Participants will be recruited for wrist assessment. They will be asked to fill out questionnaires about the functional result related to their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. All the patients suffered from traumatic or degenerative mid-carpal wrist arthritis or instability and treated surgically with arthroscopic midcarpal wrist arthrodesis in the Division of Plastic Surgery and Hand Surgery University Hospital Zürich from January 2015 to October 2017 will be included.
2. Signed informed consent for participation in the study and for further use of collected data.

Exclusion Criteria:

1. Missing Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of arthroscopic mid-carpal wrist arthrodesis for mid-carpal arthritis, related to post-traumatic or degenerative carpal deformity, performed in our Division from January 2015 to October 2017 will be studied. The approximate number of participants will be 15. There will be no control group.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Wrist range of motion after surgery | 5 minutes
  Extension , Flexion, Radial and ulnar deviation, Pronation , Supination

SECONDARY OUTCOMES:
Hand strength after surgery | 2 minutes
  Strength measurement in kilos (Kg) with Jamar Dynamometer placed in Scale 2. Three consecutive trials will be executed, the best result (higher strength in kilos) will be registered.
Pain assessment in weight bearing (Visual analogue scale, VAS) | 1 minute
  The patients will be asked to evaluate the pain in the wrist by full weight bearing, according to visual analogue scale (VAS 0-10, 0 means no pain, 10 means maximum pain)
Function assessment through DASH (The disabilities of the arm, shoulder, hand) questionnaire | 5 minutes
  This questionnaire asks about patient's symptoms as well as their ability to perform certain activities in the last week. The DASH Outcome Measure is scored in two components: the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). The response to the first 30 items of the DASH are added to form the raw, or actual, score. A minimum score is 30; a maximum is 150.The raw score is then transformed to a zero-to-100 scale with zero reflecting no disability (good function) and 100 reflecting maximum disability.
  The maximum score of the second section is 20 with a minimum of 4. The range of scores is therefore 16. This score is also transformed to a zero-to-100 scale with lower scores reflecting minimal disability, and higher scores reflecting more disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Olga Politikou, Zurich, Schweiz, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] del Pinal F, Tandioy-Delgado F. (Dry) arthroscopic partial wrist arthrodesis: tips and tricks. Handchir Mikrochir Plast Chir. 2014 Oct;46(5):300-6. doi: 10.1055/s-0034-1387707. Epub 2014 Oct 7. PMID 25290275
- [Result] del Pinal F, Klausmeyer M, Thams C, Moraleda E, Galindo C. Early experience with (dry) arthroscopic 4-corner arthrodesis: from a 4-hour operation to a tourniquet time. J Hand Surg Am. 2012 Nov;37(11):2389-99. doi: 10.1016/j.jhsa.2012.08.026. PMID 23101536